CLINICAL TRIAL: NCT00005406
Title: Change in Coronary Heart Disease Risk Factors in Young Adults
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4323; R03HL046211 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To prospectively examine changes in lipids, lipoproteins, and blood pressure among 295 young adults who had been followed for sixteen years in the Beaver County Lipid Study. The Beaver County Lipid Study tracked the cholesterol values of 295 children, ages 11 to 14 at baseline.

DETAILED DESCRIPTION:
BACKGROUND:

Epidemiologic studies of coronary risk factors have been performed primarily in populations of middle-aged adults, children, and adolescents. Relatively little is known about these risk factors in men and women 20-29 years of age.

This study provided important insights into the determinants of coronary heart disease risk factors in young adults and bolstered the argument of those who favor the early identification of and intervention in the young coronary candidate.

DESIGN NARRATIVE:

Three cross-sectional examinations had been carried out: 1) 1972-1973; 2) 1980-1981; and 3) 1988-1989. The study examined the predictors of change in total cholesterol (from examination 1 to examination 3, and change in LDL-C, HDL-C, and triglycerides between examinations 2 and 3. It also investigated the stability in several health habits and behaviors such as cigarette smoking, alcohol use, adherence to a low fat/low cholesterol diet, and physical activity. Weight gain and oral contraceptive use had been shown in previous analyses to be strong predictors of several lipids and lipoproteins.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-05; Study Completion 1992-04 (Actual)